CLINICAL TRIAL: NCT01286220
Title: A Randomized, Controlled, Evaluator-blinded Study to Evaluate the Efficacy of Dilute Bleach Baths on Skin Disease Control in Pediatric Patients With Atopic Dermatitis
Brief Title: Dilute Bleach Baths in Pediatric Patients With Atopic Dermatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study was terminated due to participant drop out
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Children's Medical Center Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 012010-059
Record Dates: First submitted 2011-01-26; First posted 2011-01-31 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Moderate to Severe Atopic Dermatitis
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dilute bleach baths (Active Comparator): Patients in the intervention group will be instructed to bathe in a dilute bleach bath twice weekly for 10 minutes.
  Interventions: Other: Dilute bleach baths
- Water (Placebo Comparator): Patients in the placebo group will be instructed to bathe in plain water twice weekly for 10 minutes.
  Interventions: Other: Water

INTERVENTIONS:
Other: Dilute bleach baths — Patients in the intervention group will be instructed to bathe in a dilute bleach bath twice weekly for 10 minutes.
  Arms: Dilute bleach baths
Other: Water — Patients in the placebo group will be instructed to bathe in plain water twice weekly for 10 minutes.
  Arms: Water

SUMMARY:
The purpose of this study is to determine if twice weekly 10 minute dilute bleach baths decreases disease severity in patients with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* 2-17 years of age at time of consent. A parent or legal guardian will be required to consent and authorize their enrollment in the study.
* Male or female of any ethnic background.
* English or Spanish speaking.
* A clinical diagnosis of atopic dermatitis for at least 6 months prior to enrollment.
* Must have moderate to severe atopic dermatitis as rated by the EASI score.
* Able to adhere to study visit schedule and other protocol requirements.
* Patients and/or family members must agree to not use any other prescription or over the counter medications other than the ones prescribed by the study protocol.

Exclusion Criteria:

* Clinical evidence of bacterial or viral superinfection on first visit.
* Have received phototherapy within 2 months prior to enrollment.
* Have received any systemic medication for atopic dermatitis or any that may affect evaluation of atopic dermatitis within 2 months prior to enrollment.
* Have a known hypersensitivity response, including anaphylaxis, to any of the topicals used for treatment (i.e. topical steroids, bleach)
* Participation in another clinical trial using an investigational agent or procedure.
* Pregnant or planning pregnancy or surgery during the participation in the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index Score (EASI) | Change in EASI score from baseline at 1 month and 3 month follow ups
  EASI score is recorded at baseline, 1 month and 3 month follow ups.

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) | Change in IGA score from baseline at 1 month and 3month follow ups
  IGA scores are recorded at baseline, 1 month and 3 month follow ups.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center of Dallas, Dallas, Texas, United States

REFERENCES:
- [Result] Huang JT, Abrams M, Tlougan B, Rademaker A, Paller AS. Treatment of Staphylococcus aureus colonization in atopic dermatitis decreases disease severity. Pediatrics. 2009 May;123(5):e808-14. doi: 10.1542/peds.2008-2217. PMID 19403473